CLINICAL TRIAL: NCT04323228
Title: Anti-inflammatory/Antioxidant Oral Nutrition Supplementation on the Cytokine Storm and Progression of COVID-19: A Randomized Controlled Trial
Brief Title: Anti-inflammatory/Antioxidant Oral Nutrition Supplementation in COVID-19
Acronym: ONSCOVID19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Mahmoud Abulmeaty, M.D., FACN., Associate Professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ONS_COVID-19
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
Keywords: COVID-19; Antioxidant ONS; Cytokine storm
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — Antioxidants

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated into two study groups; intervention group (IG, n=20) and placebo group (PG, n=20). Computer-generated random numbers will be used to randomize the participants into one of two intervention groups.
Who Masked: Participant, Care Provider
Masking Description: The intervention-supplement and isocaloric-placebo will be served in the same shape, size and color. the care providers (nurses, dietitians) will not know members of each groups or the nature or composition of the ONS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): the intervention groups will receive daily oral antioxidant supplement enriched in vitamin A, C, E, Selenium and Zinc. The composition of one capsule of the intervention-supplement includes: 1500 mcg vitamin A (as β-carotene), 250 mg Vitamin C, 90 mg vitamin E, 15 ug Selenium, and 7.5 mg Zinc.
  Interventions: Dietary Supplement: Oral supplement enriched in antioxidants
- Placebo (Placebo Comparator): Placebo group will receive daily intervention in form of cellulose-containing gelatin capsules with the same color and shape.
  Interventions: Dietary Supplement: cellulose-containing placebo capsules

INTERVENTIONS:
Dietary Supplement: Oral supplement enriched in antioxidants — the intervention group will receive a commercially available antioxidant supplement, which will be given to patients with COVID-19 in the morning after breakfast.
  Arms: Intervention
Dietary Supplement: cellulose-containing placebo capsules — The placebo group will receive an oral supplement at the same time in the same shape/size/color.
  Arms: Placebo

SUMMARY:
COVID-19 pandemic threatens patients, societies and healthcare systems around the world. The host immunity determines the progress of the disease and its lethality. The associated cytokine storm mainly affects the lungs; leading to acute lung injury with variable degrees. Modulation of cytokine production using Immunonutrition is a novel concept that has been applied to other diseases. Using specific nutrients such as n3- fatty acids and antioxidant vitamins in extraordinary doses modulate the host immune response and ameliorate the cytokine storm associated with viral diseases such as COVID-19. In this proposal, we will conduct a prospective double-blinded controlled trial for 14 days on 30 SARS-CoV-2 positive cases. The participant will be randomly assigned to two groups (n=20/each); intervention (IG) and placebo (PG) groups. The IG group will be provided with an anti-inflammatory and antioxidant oral supplement (OS) on a daily basis, while the PG will be given an isocaloric placebo. Basal and weekly nutritional screening, as well as recording of anthropometric, clinical and biochemical parameters, will be done. The main biochemical parameters include serum ferritin level, cytokine storm parameters (interleukin-6, Tumor necrosis factor-α, and monocyte chemoattractant protein 1), C-reactive protein, total leukocyte count, differential lymphocytic count and neutrophil to lymphocyte ratio. It is expected that the anti-inflammatory-antioxidant OS might help in the reduction of the COVID-19 severity with more preservation of the nutritional status of infected cases.

DETAILED DESCRIPTION:
Subjects: A total of 40 participants will be enrolled in this double-blinded prospective, randomized controlled trial. All participants will sign a written consent after details of the study have been fully explained to them. Later on, they will be randomly allocated into two study groups; intervention group (IG, n=20) and placebo group (PG, n=20). Computer-generated random numbers will be used to randomize the participants into one of two intervention groups. The study protocol will be approved by the IRB committee in King Khalid University Hospital, King Saud University Medical city. This clinical trial will be registered in the clinicaltrials.gov registry.

Settings: All participants will be SARS-CoV-2 positive cases admitted to King Khalid University Hospital.

Study protocol: All study participants will be instructed to either consume one capsule of oral supplement enriched in antioxidants vitamins or placebo. The OS will be served in opaque capsules of the same size, shape and color and should be ingested in the morning under the supervision of a nurse. The OS should not be consumed before the time of a meal. The composition of one capsule of the intervention-OS includes: enriched in vitamin A, C, E, Selenium and Zinc. The composition of one capsule of the intervention-supplement includes: 1500 mcg vitamin A (as β-carotene), 250 mg Vitamin C, 90 mg vitamin E, 15 ug Selenium, and 7.5 mg Zinc. The composition of the placebo will have the same weight of cellulose, and zero concentrations of vitamin A, C, E, Selenium and zinc.

All participants will be assessed at the start and reassessed again after 1 week and after 14-days period. The assessment will include nutritional screening by Nutritional risk screening 2002 (NRS-2002), Subjective global assessment (SGA), and Global Leadership Initiative on Malnutrition (GLIM) criteria. Besides anthropometric measures, clinical Global Leadership Initiative on Malnutrition (GLIM). also, anthropometric measurements, clinical assessment, and biochemical data will be measured. Statistical analysis: The Statistical Package for the Social Sciences (SPSS) version 25 will be used for analysis. The descriptive statistics for continuous variables will be presented as mean ± standard deviation, while other categorical variables as percentages. The independent sample t-test will be used for comparison between the IG and PG groups. For repeated measures at multiple points of time will be tested by Friedman's two-way ANOVA. The Pearson correlation coefficient will be applied to correlate some relevant variables. All these tests were performed with 80% power and a 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV-2 infection
* COVID-19 patient in stable condition (i.e., not requiring ICU admission).

Exclusion Criteria:

* Tube feeding or parenteral nutrition.
* Pregnant or lactating women
* Admission to ICU > 24 hours
* participation in another study including any forms of supplementation or disease specific ONS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline score of Nutrition risk screening-2002 (NRS-2002) at end of the trial | up to 3 months
  Changes in scores of the NRS-2002 for patients with COVID-19 at the end of the study, from 0 to 7 scores, with those scores < 3 means no risk of malnutrition and >= 3 means malnutrition.
Change from baseline Serum ferritin level at end of the trial | up to 3 months
  Change in serum ferritin at the end of the trial as ferritin is considered as a COVID-19 fatality predictor.
Change from baseline serum Interleukin-6 concentration at end of the trial | up to 3 months
  Change in IL-6 at the end of the trial as it represent the cytokine storm and it is considered as a COVID-19 fatality predictor
Change from baseline serum C-reactive protein concentration at end of the trial | up to 3 months
  Change in C-reactive protein in the serum at the end of the trial which reflect the acute phase
Change from baseline serum Tumor necrosis factor-α concentration at end of the trial | up to 3 months
  Change in the TNF a in the serum at the end of study as it represent severity of the cytokine storm
Change from baseline serum monocyte chemoattractant protein 1 (MCP-1) at end of the trial | up to 3 months
  plasma MCP-1 represent severity of the cytokine storm

SECONDARY OUTCOMES:
Change from baseline Weight at end of the trial | up to 3 months
  Body weight in Kg
Height | up to 1 month
  stature in cm
Change from baseline BMI at end of the trial | up to 3 months
  Claculation of BMI according to weight / square Height
Change from baseline mid arm circumference at end of the trial | up to 3 months
  changes of MAC in cm
Change from baseline triceps skin-fold thickness at end of the trial | up to 3 months
  changes of TSF in mm
Change from baseline MAMA at end of the trial | Up to 3 months
  ). The mid-arm muscle area (MAMA) will be calculated according to the following equation: {MAMA= (MAC - π x TSF)2 / 4π}.
Change from baseline percentage of peripheral O2 saturation at end of the trial | up to 3 months
  changes in the percentage of peripheral O2 saturation by an oximeter
Change from baseline degree of body temperature at end of the trial | up to 3 months
  changes in the degree of body temperature by infrared thermometer
Change from baseline count the total leukocyte at end of the trial | up to 3 months
  change in the count from complete blood counts
Change from baseline differential lymphocytic count at end of the trial | up to 3 months
  change in the count from complete blood counts
Change from baseline Neutrophil count at end of the trial | up to 3 months
  change in the count from complete blood counts
Change from baseline neutrophil to lymphocyte ratio at end of the trial | up to 3 months
  change in the rations calculated by division of the neutrophil count by the lymphocyte count

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Mohamed BinAbdulaziz Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication.
Access Criteria: Access will be available for any researcher interested in this type of research on considerable consent.

REFERENCES:
- [Background] Abulmeaty MM, Almajwal AM, Almadani NK, Aldosari MS, Alnajim AA, Ali SB, Hassan HM, Elkatawy HA. Anthropometric and central obesity indices as predictors of long-term cardiometabolic risk among Saudi young and middle-aged men and women. Saudi Med J. 2017 Apr;38(4):372-380. doi: 10.15537/smj.2017.4.18758. PMID 28397943
- [Background] Grimm H, Calder PC. Immunonutrition. Br J Nutr. 2002 Jan;87 Suppl 1:S1. doi: 10.1079/bjn2001450. No abstract available. PMID 11895145
- [Background] Calder PC. Immunonutrition in surgical and critically ill patients. Br J Nutr. 2007 Oct;98 Suppl 1:S133-9. doi: 10.1017/S0007114507832909. PMID 17922951
- [Background] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360
- [Background] Das SK, Chisti MJ, Sarker MHR, Das J, Ahmed S, Shahunja KM, Nahar S, Gibbons N, Ahmed T, Faruque ASG, Rahman M, J Fuchs G 3rd, Al Mamun A, John Baker P. Long-term impact of changing childhood malnutrition on rotavirus diarrhoea: Two decades of adjusted association with climate and socio-demographic factors from urban Bangladesh. PLoS One. 2017 Sep 6;12(9):e0179418. doi: 10.1371/journal.pone.0179418. eCollection 2017. PMID 28877163
- [Background] Harada K, Minami H, Ferdous T, Kato Y, Umeda H, Horinaga D, Uchida K, Park SC, Hanazawa H, Takahashi S, Ohota M, Matsumoto H, Maruta J, Kakutani H, Aritomi S, Shibuya K, Mishima K. The Elental(R) elemental diet for chemoradiotherapy-induced oral mucositis: A prospective study in patients with oral squamous cell carcinoma. Mol Clin Oncol. 2019 Jan;10(1):159-167. doi: 10.3892/mco.2018.1769. Epub 2018 Nov 16. PMID 30655992
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Kim H. Glutamine as an immunonutrient. Yonsei Med J. 2011 Nov;52(6):892-7. doi: 10.3349/ymj.2011.52.6.892. PMID 22028151
- [Background] Kondrup J, Allison SP, Elia M, Vellas B, Plauth M; Educational and Clinical Practice Committee, European Society of Parenteral and Enteral Nutrition (ESPEN). ESPEN guidelines for nutrition screening 2002. Clin Nutr. 2003 Aug;22(4):415-21. doi: 10.1016/s0261-5614(03)00098-0. PMID 12880610
- [Background] McCowen KC, Bistrian BR. Immunonutrition: problematic or problem solving? Am J Clin Nutr. 2003 Apr;77(4):764-70. doi: 10.1093/ajcn/77.4.764. PMID 12663270
- [Background] Mariette C. Immunonutrition. J Visc Surg. 2015 Aug;152 Suppl 1:S14-7. doi: 10.1016/S1878-7886(15)30005-9. PMID 26315574
- [Background] McCarthy MS, Martindale RG. Immunonutrition in Critical Illness: What Is the Role? Nutr Clin Pract. 2018 Jun;33(3):348-358. doi: 10.1002/ncp.10102. PMID 29878555
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Tisoncik JR, Korth MJ, Simmons CP, Farrar J, Martin TR, Katze MG. Into the eye of the cytokine storm. Microbiol Mol Biol Rev. 2012 Mar;76(1):16-32. doi: 10.1128/MMBR.05015-11. PMID 22390970
- [Background] Teo BW, Toh QC, Chan XW, Xu H, Li JL, Lee EJ. Assessment of muscle mass and its association with protein intake in a multi-ethnic Asian population: relevance in chronic kidney disease. Asia Pac J Clin Nutr. 2014;23(4):619-25. doi: 10.6133/apjcn.2014.23.4.01. PMID 25516320
- See also: Immunonutrition: Interactions of Diet, Genetics, and Inflammation - Google Books. In Immunonutrition: Interactions of Diet, Genetics, and Inflammation — https://books.google.com.sa/books?id=d2HvAgAAQBAJ&pg=PA17&lpg=PA17&dq=immunonutrition+virus&source=bl&ots=VUneSrxucb&sig=ACfU3U0bKU0mAdShOEvzIAMifj7SNE47Lw&hl=en&sa=X&redir_esc=y#v=onepage&q=immunonutrition%20virus&f=false